CLINICAL TRIAL: NCT06233188
Title: Does the Patient-specific Depth of the Lateral Nasal Wall Osteotomy Affect the Pterygomaxillary Separation During le Fort I Down-fracture?
Brief Title: Effect of Customized Lateral Nasal Wall Osteotomy on the Pterygomaxillary Separation During le Fort I Down-fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Taha Pergel, Assistant Profesor, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-E.110541
Record Dates: First submitted 2024-01-10; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Malocclusion; Open Bite; Le Fort; I; Orthognathic Surgery
Keywords: orthognatic surgery; le fort I; arterial bleeding; down fracture; lateral nasal wall; pterygomaxillary junction
MeSH Terms: conditions — Malocclusion; Open Bite

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): In the study group, lateral nasal osteotomy was performed 2 mm less than the measured distance in the axial section
  Interventions: Procedure: orthogantic surgery
- conventional group (Active Comparator): n the conventional osteotomy group, lateral nasal osteotomy was performed 25 mm for female and 30 mm for male patients, as suggested in the literature.
  Interventions: Procedure: orthogantic surgery

INTERVENTIONS:
Procedure: orthogantic surgery — surgery that correcting the maxilla and mandible related with each other

SUMMARY:
The goal of this clinical trial is to show the effect of patient specific lateral nasal wall osteotomy to the pterygomaxillary separation during Le Fort I down-fracture.

Participants will be divided into two treatment groups. In study group, surgery planned according to the patients' indivudial anatomy and in the conventional group, surgery planned according to mean anatomical datas.

Researchers will compare patient specific lateral nasal wall osteotomy to see if it affects the pterygomaxillary junction seperation during le fort I downfracture.

DETAILED DESCRIPTION:
The same surgical team performed the osteotomies under general anesthesia with nasotracheal intubation. Hypotensive anesthesia was applied as a standard protocol in all patients. Orthognathic surgery, including Le Fort I and sagittal split ramus osteotomy, was used to correct skeletal deformities.

Bone osteotomy was initiated on the bilateral wall of the maxilla with piezosurgery after a mucosal incision and flap elevation.Lateral nasal osteotomy (LNO) with Nievert Anderson single guarded osteotome, median septum separation with double guarded U-shaped osteotome, and pterygomaxillary junction separation with curved osteotome were performed before the down-fracture. The only difference between the conventional and study groups was the depth of the LNO. In the study group, LNO was performed at a depth of 2 mm less than the measured distance in the axial section. In the conventional osteotomy group, LNO was performed at 30 mm for females and 35 mm for males, as suggested in the literature. A curved osteotome and a mallet were used in each case to separate the pterygomaxillary junction. The down-fracture of the maxilla was performed using a hook and a bone spreader in all patients. When the maxilla was down-fractured, LNW and the pterygomaxillary separation types were assessed intraoperatively. The maxilla was stabilized in its new position by four L-shaped osteosynthesis mini-plates at the zygomaticomaxillary buttress and the aperture piriformis regions.

ELIGIBILITY:
Inclusion Criteria: The inclusion criteria

* orthognathic surgery to treat malocclusion
* sleep apnea
* jaw asymmetry

Exclusion Criteria:

* cleft lip and palate
* previous orthognathic surgery
* rhinoplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
lateral nasal wall separation | 1 year
  The primary outcome variable is lateral nasal wall separation:
  Type 1 Separation from the osteotomy line
  Type 2 Separation 2-4 mm above the osteotomy line
  Type 3 Separation 4 mm or more above the osteotomy line

SECONDARY OUTCOMES:
pterygomaxillary junction separation | 1 year
  The secondary outcome variable is pterygomaxillary separation
  Type 1 Separation including the tuber maxilla
  Type 2 Separation from the pterygomaxillary junction
  Type 3 Separation including the pterygoid plates

CONTACTS AND LOCATIONS:
Locations (1):
- Taha Pergel, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided